CLINICAL TRIAL: NCT04809844
Title: Retrospective Study of Concurrent Paclitaxel and Radiation Therapy After Adjuvant Doxorubicin and Cyclophosphamide Chemotherapy for Stage 2 or 3 Breast Cancer
Brief Title: Concurrent Paclitaxel and Radiotherapy After Adjuvant Doxorubicin and Cyclophosphamide for Stage 2 or 3 Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hoda Gamal Boraey, Principal investigator, Assiut University
Other Study IDs: Breast cancer in females
Record Dates: First submitted 2021-03-13; First posted 2021-03-22 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Concurrent chemoradiation — concurrent Paclitaxel and radiation therapy after Adjuvant doxorubicin and Cyclophosphamide chemotherapy for stage ll or lll breast cancer .

SUMMARY:
The aim of this study is Evaluation of the efficacy & toxicity of concurrent paclitaxel and breast radiotherapy and assesment of overall survival & progression free survival

DETAILED DESCRIPTION:
Over the recent years , breast cancer remains the most common cancer in women in the world . With nearly 107 Million new Cases diagnosed in 2012 (second most common cancer over all) . this represent about 12 % of all new cancer cases and 25 % of all cancers in women . By contrast the mortality rate has declined dramatically since the introduction of adjuvant systemic therapy & radiation therapy, which are now used extensively for their established benefit in local (radiotherapy ) ,survival without metastasis (chemotherapy) and overall survival of both of them . However , the optimal sequence of chemotherapy & radiotherapy remain controversial three sequence were investigated:

1. Delivering all radiotherapy first .
2. A " Sandwich " approach .
3. Delivering all chemotherapy first . Observational studies have suggested that delaying initiation of chemotherapy increase the incidence of distant metastasis & delaying the initiation therapy more than 6 months after breast cancer diagnosis might increase risk of local regional recurrence . Concurrent chemoradiation therapy has an advantage of shortening the duration of therapy , allowing radiotherapy & chemotherapy to start temporally and potentially improving local control via radiation sensitizing effect of chemotherapy.The feasibility of concurrent radiotherapy with taxane, which constitute a standard treatment used as adjuvant therapy has been evaluated in stage II,III breast cancer. Taxane Promote stabilization of microtubules causing cell cycle arrest in G2/M junction and serve as radio sensitizing agents.In a prospective study using Paclitaxel & radiotherapy concurrently Paclitaxel given every 3 weeks for 4 cycles the authors concluded that Concurrent chemoradiation therapy improve local control with acceptable toxicity.

ELIGIBILITY:
Inclusion criteria :

* • This study will include women aged 18 years &older.
* patients must be histologically diagnosed with breast cancer (ductal & others).
* patients who underwent conservative breast surgery & modified radical mastectomy.
* patients with stage ll&lll breast cancer.
* patients who received (AC) as adjuvant treatment .

Exclusion Criteria:

* patients with stage 1 or 4 breast cancer.
* patients received adjuvant chemotherapy rather than (AC) .
* patients with prior irradiation with thoracic region .
* pregnancy or lactation .
* patient with serious comorbid disease such as chronic obstructive pulmonary disease .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study will include female patients with stage II-lll breast cancer who underwent conservative breast surgery & modified radical mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity of concurrent paclitaxel & breast radiotherapy such as acute skin toxicities . | baseline
  Acute skin toxicities will be graded by using a scale ranging from 0-4 where 0= no change ,1= follicular, faint or dull erythema/epilation/ dry desquamation , 2= tender or bright erythema , 3= confluent moist desquamation , pitting edema , 4= ulceration , hemorrhage , necrosis .

REFERENCES:
- [Background] Ghoncheh M, Pournamdar Z, Salehiniya H. Incidence and Mortality and Epidemiology of Breast Cancer in the World. Asian Pac J Cancer Prev. 2016;17(S3):43-6. doi: 10.7314/apjcp.2016.17.s3.43. PMID 27165206
- [Background] Olivotto IA, Bajdik CD, Plenderleith IH, Coppin CM, Gelmon KA, Jackson SM, Ragaz J, Wilson KS, Worth A. Adjuvant systemic therapy and survival after breast cancer. N Engl J Med. 1994 Mar 24;330(12):805-10. doi: 10.1056/NEJM199403243301201. PMID 8114832
- [Background] Abal M, Andreu JM, Barasoain I. Taxanes: microtubule and centrosome targets, and cell cycle dependent mechanisms of action. Curr Cancer Drug Targets. 2003 Jun;3(3):193-203. doi: 10.2174/1568009033481967. PMID 12769688
- [Background] Ali Hassan A, Ibrahim NY, Jassen MAR. Concurrent Paclitaxel and Radiotherapy for Node Positive Breast Cancer. Gulf J Oncolog. 2019 Jan;1(29):14-21. PMID 30956192